CLINICAL TRIAL: NCT02511223
Title: PHASE II Study - EFFICACY AND SAFETY OF (PARPi )Polyadenosine Diphosphoribose [Poly Polymerisation inhibitorTO TREAT PANCREATIC CANCER
Brief Title: Efficacy and Safety of PARPi to Treat Pancreatic Cancer
Acronym: 10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-14-2358-TG-CTIL
Record Dates: First submitted 2015-07-01; First posted 2015-07-29 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Only one Arm,All patients will receive Olaparib 300 (mg) milligram bid p.o till disease progression
  Interventions: Drug: OLAPARIB

INTERVENTIONS:
Drug: OLAPARIB — Olaparib 300 (mg) twice a day per os given every day until disease progression or toxicity
  Other Names: PARPi

SUMMARY:
This is an open label, single arm, phase II trial of Olaparib for (PDAC) pancreatic ductal adenocarcinoma patients with BRCAness (breast cancer gene). All study subjects will receive Olaparib in a dose of 300 mg p.o twice daily. Treatment will continue until progression, intolerable toxicity or as per patient preference.

Primary objective:

To determine the efficacy of Olaparib monotherapy in stage IV pancreatic ductal adenocarcinoma (PDAC)with (BRCAness) BRCA -Breast Cancer susceptibility gene.

DETAILED DESCRIPTION:
An open label, single arm, phase II trial of Olaparib for PDAC patients with BRCAness (BRCA-Breast Cancer susceptibility gene).

Patients with previously identified Loss of ATM (ATM serine/threonine kinase)by (IHC) Immunohistochemistry OR (overall survival) - Family history of BRCA (Brest Cancer gene)-associated cancers: breast, ovarian, pancreatic, gastric or prostate must be present in 2 or more first-degree relatives OR- Patients with previously identified genetic aberrations that are associated with (HRD) Homologous recombination deficiency will be eligible [e.g. somatic BRCA mutation, Fanconi Anemia gene or RAD51(eukaryote gene) mutations].

All patients will be retrospectively investigated for (HRD)Homologous recombination repair deficiencies signature using transcriptome profiling and ATM expression and the results correlated with (PARPi) (Polyadenosine 5'diphosphoribose [poly (ADP ribose)] polymerization INHIBITOR) response rates.

Eligible patients will receive treatment with Olaparib tablets p.o 300 (mg) milligram twice daily until progression. Each treatment cycle is described as 28 days long. Patients will have tumor assessments according to RECIST 1.1(Response Evaluation Criteria In Solid Tumors) at baseline. Patients will then be followed for the final analysis of (OS) overall survival.

Eligible patients will be those patients with stage IV pancreas cancer previously treated for metastatic disease. Patients must have received one prior therapy for the treatment of metastatic disease or refused chemotherapy.

Following study entry, patients will attend clinic visits every two weeks for the first 4 weeks of treatment (Days 1 and 15,). Patients will then attend clinic visits every 4 weeks whilst on study treatment.

Patients should continue to receive study treatment until objective radiological disease progression as per RECIST as assessed by the investigator and as long as in the investigator's opinion they are benefiting from treatment and they do not meet any other discontinuation criteria.

Following discontinuation of study treatment, patients should be seen at 30 days post discontinuation for the evaluations outlined in the study schedule. Patients will be contacted in the 7 days following a specified date (data cut-off date) to capture survival status at that point for each survival analysis.

Patients will have tumor assessments according to RECIST at baseline and every 8 weeks (±1week) up to 40 weeks and then every 12 weeks (±1 week) relative to date of enrolment until objective radiological disease progression according to modified RECIST criteria. Ongoing collection of site review tumor assessment is required and must be recorded in the electronic case report form (eCRF).

Any patient who discontinues study treatment for reasons other than objective radiological progression should continue to undergo scheduled objective tumor assessments according to the study schedule, in order to assess objective radiological progression of disease. Failure to do so may result in bias to the study results.

ELIGIBILITY:
Inclusion Criteria:

* • Patients must be male or female ≥18 years of age

  * Patients with histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas.
  * Patients must have tested negative for BRCA 1 or 2 germline deleterious mutation or be ineligible for BRCA testing [as determined by their insurer]
  * Patients with previously identified Loss of ATM by IHC OR
  * Family history of BRCA-associated cancers: breast, ovarian, pancreatic, gastric or prostate must be present in 2 or more first-degree relatives OR
  * Patients with previously identified genetic aberrations that are associated with HRD will be eligible [e.g. somatic BRCA mutation, Fanconi Anemia gene or RAD51 mutations].
  * Patients must have received at least one prior therapy for metastatic disease or have refused chemotherapy to be eligible
  * Patients with measurable disease and/or non-measurable or no evidence of disease assessed at baseline by CT (or MRI where CT is contraindicated) will be entered in this study. RECIST 1.1 has been modified to allow the assessment of progression due to new lesions in patients with no evidence of disease at baseline
  * (ECOG) Eastern Cooperative Oncology Group: A performance status using scales and criteria to assess how a patient's disease is progressing)Performance Status 0-1 (Karnofsky >70).
  * Patients must have adequate organ and marrow function as defined below:
* Leukocytes >3,000 cells/mm3
* Absolute neutrophil count >1,500 cells/mm3
* Platelets >100,000 cells/mm3
* Hemoglobin >9 g/dl (no blood transfusions within 4 weeks prior to enrolment)
* Total bilirubin <1.5 X institutional upper limit of normal (IULN)
* (AST) aspartate aminotransferase (SGOT)/(ALT) Alanine transaminase(SGPT) <2.5 X IULN without liver metastasis <5 X IULN for patients with liver metastasis
* Creatinine within normal institutional limits OR
* Creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal

  * (INR)international normalized ratio <1.5
  * Women of childbearing potential (defined as not post-menopausal for 12 months or no previous surgical sterilization) and fertile men must agree to use adequate contraception for the duration of study participation. Male subjects must agree to refrain from sperm donation during the study and for 30 days after the last dose of study drugs.
  * Ability to understand and the willingness to sign a written informed consent document. Signed informed consent form must be obtained prior to initiation of study evaluations and/or activities.

Exclusion Criteria:

* Uncontrolled intercurrent illness including symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia and myocardial infarction (MI) within 3 months of initiation of therapy.

  * Pregnancy or lactation
  * Patient has active and uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
  * Patient has undergone major surgical resection within 4 weeks prior to enrollment.
  * Patient received radiotherapy, surgery, chemotherapy, or an investigational therapy within 2 weeks prior to study entry.
  * Patient has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug
  * Serious psychiatric or medical conditions that could interfere with treatment
  * History of prior malignancy unless the malignancy has been treated with no evidence of active disease and more than 2 years from initial diagnosis
  * Major bleeding in the last 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by using RECIST 1.1 | approximately- 24 months
  Due to lack of results, study has been early terminated

CONTACTS AND LOCATIONS:
Overall Officials: Talia Golan, MD, Principal Investigator — Sheba Medical Centre, Israel
Locations (1):
- Sheba Medical Centre, Ramat Gan, Israel